CLINICAL TRIAL: NCT04130490
Title: The Heidelberg Engineering ANTERION Anterior Segment Cornea and IOL Precision and Agreement Study
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B-2018-5
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cataract; Healthy Eye; Cornea Abnormality; Post-Keratorefractive Surgery; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Eye with normal Anterior Segment: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION
- Eye with cataract: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION
- Eye with corneal abnormality: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION
- Eye with status post-keratorefractive surgery: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION
- Eye without a crystalline lens: 3 repeat measurements on each of the 3 investigational and reference devices
  Interventions: Device: ANTERION

INTERVENTIONS:
Device: ANTERION — 3 repeat measurements performed with two of the ANTERION acquisition types and 3 repeat measurements performed with 2 acquisition types of the references devices

SUMMARY:
This is a prospective clinical study that will be conducted at one clinical site located in the United States to assess anterior segment parameters with the ANTERION

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 years or older
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions
3. Able to fixate
4. With the following eye pathology status for the individual eye population:

   * A. Eye with normal anterior segment and crystalline lens
   * B. Eye with a cataract of grade 1.5 or higher
   * C. Eye with abnormal corneal shape
   * D. Eye with status post-keratorefractive surgery
   * E. Eye without a crystalline lens

Exclusion Criteria:

1. Subjects which were enrolled in the B-2018-1 clinical study
2. Active infection or inflammation in the study eye
3. Insufficient tear film or corneal reflex
4. Physical inability to be properly positioned at the study devices or eye exam equipment
5. Rigid contact lens wear 2 weeks prior to imaging
6. Soft lenses worn within one hour prior to imaging
7. With the following eye pathology status for the individual eye population:

   * A. Eye meets eligibility criteria for eye populations B, C, D or E
   * B. Eye meets eligibility criteria for eye populations C,D or E
   * C. Eye meets eligibility criteria for eye populations D or E
   * E. Eye with abnormal corneal shape (except status post-keratorefractive surgery)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eyes with normal anterior segment and crystalline lens; eyes with cataract of grade 1.5 or higher; eyes with abnormal corneal shape; eyes with status post-keratorefractive surgery and eyes without a crystalline lens
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Precision and Agreement 1 | 1 day
  Reproducibility, repeatability and agreement of Anterior Corneal Topography parameters (3mm ring) of ANTERION and the reference device
Precision and Agreement 2 | 1 day
  Reproducibility, repeatability and agreement of Anterior Corneal Topography parameters (6mm zone) of ANTERION and the reference device
Precision and Agreement 3 | 1 day
  Reproducibility, repeatability and agreement of Posterior Corneal Topography parameters (3mm ring) of ANTERION and the reference device
Precision and Agreement 4 | 1 day
  Reproducibility, repeatability and agreement of Posterior Corneal Topography parameters (6mm zone) of ANTERION and the reference device
Precision and Agreement 5 | 1 day
  Reproducibility, repeatability and agreement of Cornea Thickness (µm) of ANTERION and the reference device
Precision and Agreement 6 | 1 day
  Reproducibility, repeatability and agreement of Lens Thickness, ACD, Pupil Diameter, White-to-White, Axial Length (mm) of ANTERION and the reference device
Precision and Agreement 7 | 1 day
  Reproducibility, repeatability and agreement of Anterior Chamber Volume (mm^3) of ANTERION and the reference device

SECONDARY OUTCOMES:
Adverse Events Rate | 1 day
  Adverse events found during the clinical study

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Dul, Principal Investigator — State University of New York College of Optometry
Locations (1):
- State University of New York College of Optometry, New York, New York, United States